CLINICAL TRIAL: NCT04733573
Title: Pressure Algometry Evaluation of Two Occlusal Splint Designs in Bruxism Management - Randomized, Controlled Clinical Trial
Brief Title: Pressure Algometry Evaluation of Two Occlusal Splint Designs in Bruxism Management - RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Dalewski Bartosz, DMD, PhD, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KB-0012/49/10
Record Dates: First submitted 2021-01-26; First posted 2021-02-02 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Bruxism; Sleep Disorder
Keywords: bruxism; algometer; pressure pain threshold; occlusal; splint; grinding; clenching
MeSH Terms: conditions — Bruxism; Sleep Wake Disorders; Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusal appliance by Okeson with canone guidance (Active Comparator): Occlusal appliance will be used while sleeping for 30 days.
  Interventions: Device: Two different occlusal splints
- Bimaxillary splint without canine guidance (Active Comparator): Bimaxillary splint will be used while sleeping for 30 days.
  Interventions: Device: Two different occlusal splints

INTERVENTIONS:
Device: Two different occlusal splints — Two different occlusal splints will be used for bruxism management, PPT would be evaluated twice - before and after 30 days of splint therapy using pressure algometer (FPX25, Wagner Instruments, US)

SUMMARY:
During the study, designated pressure points before and after one month of splint usage will be evaluated as possible indicators of two different splints efficacy..

Two study groups will be formed. The study will be conducted on patients reporting to the Dental Prosthetics Outpatient Clinic of PUM in Szczecin, Poland. Patients aged 18-65 years with probable bruxism, yet requiring splint therapy will be included in the study.

DETAILED DESCRIPTION:
During the study, designated pressure points before and after one month of splint usage will be evaluated as possible indicators of two different splints efficacy..

Two study groups will be formed. The study will be conducted on patients reporting to the Dental Prosthetics Outpatient Clinic of PUM in Szczecin, Poland. Patients aged 18-65 years with probable bruxism, yet requiring splint therapy will be included in the study. Probable bruxism will be diagnosed on the basis of the patient's history and examination as follows. Inclusion criteria:

I. Nocturnal Bruxism according to International Classification of Sleep Disorders, Second Edition (ICSD-2).

A. The patient reports or is aware of tooth-grinding sounds or tooth clenching during sleep.

B. One or more of the following is present: a. Abnormal wear of teeth b. Jaw muscle discomfort, fatigue, or pain and jaw lock upon awakening. c. Masseter muscle hypertrophy upon voluntary forceful clenching.

C. The jaw muscle activity is not better explained by another current sleep disorder, medical or neurological disorder, medication use, or substance use disorder.

II. Additional questionnaire for detecting bruxers:

1. Has anyone heard you grinding your teeth at night?
2. Is your jaw ever fatigued or sore in the morning?
3. Are your teeth or gums ever sore on awakening in the morning?
4. Do you ever experience temporal headaches on awakening in the morning?
5. Are you aware of grinding your teeth during the day?
6. Are you ever aware of clenching your teeth during the day
7. Can you imitate a sound of grinding using your teeth.

III. Eligible patients will be randomly assigned into two groups. Sealed, opaque envelopes will be used for randomization. The first group will be treated with a stabilization appliance described by Okeson. The second group will undergo therapy with a two-jaw splint with an arch. Patients will be informed about how to use and maintain hygiene of the splint. It will be recommended to use a splint only while sleeping.

IV. Pressure pain threshold test (PPT) will be carried out at the Department of Prosthodontics of the Pomeranian Medical University, Szczecin, Poland using the Wagner Paintest FPX 25 algometer. Points within the following muscles will be examined:

masseter muscles, anterior, middle and posterior abdomens of the temporal muscles, a point at the height of the TMJ larger exterior convexity, the sternocleidomastoid muscles and the preauriculare point, bilaterally two measurements at each visit. The test will be performed at the first visit and after 30 days of therapy.

The algometer comes with a 1 cm2 rubber tip, which measures the pressure in kg / s while pressing on the tested surface. Both test results will be used as a pre- and post- treatment evaluation.

ELIGIBILITY:
Inclusion Criteria:

* I. Nocturnal Bruxism according to International Classification of Sleep Disorders, Second Edition (ICSD-2).

A. The patient reports or is aware of tooth-grinding sounds or tooth clenching during sleep.

B. One or more of the following is present: a. Abnormal wear of teeth b. Jaw muscle discomfort, fatigue, or pain and jaw lock upon awakening. c. Masseter muscle hypertrophy upon voluntary forceful clenching.

C. The jaw muscle activity is not better explained by another current sleep disorder, medical or neurological disorder, medication use, or substance use disorder.

II. Additional questionnaire for detecting bruxers:

Has anyone heard you grinding your teeth at night? Is your jaw ever fatigued or sore in the morning? Are your teeth or gums ever sore on awakening in the morning? Do you ever experience temporal headaches on awakening in the morning? Are you aware of grinding your teeth during the day? Are you ever aware of clenching your teeth during the day Can you imitate a sound of grinding using your teeth.

Exclusion Criteria:

* unrestored tooth losses
* patients wearing removable dentures of any kind
* psychiatric conditions undermining/preventing occlusal splint usage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold in designated points | 30 days
  Evaluation of difference between algometer readings before and after 30 days of splint usage - FPX25 algometer (Wagner instruments, US) will be used

CONTACTS AND LOCATIONS:
Overall Officials: Agata Kamińska, DMD, Principal Investigator — Pomeranian Medical Universiy in Szczecin, Poland
Locations (1):
- Chair and Depratment of Dental Prosthetics, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dalewski B, Kaminska A, Kiczmer P, Wegrzyn K, Palka L, Janda K, Sobolewska E. Pressure Algometry Evaluation of Two Occlusal Splint Designs in Bruxism Management-Randomized, Controlled Clinical Trial. J Clin Med. 2021 May 27;10(11):2342. doi: 10.3390/jcm10112342. PMID 34071832
- See also: https://www.mdpi.com/2077-0383/10/11/2342 — https://pubmed.ncbi.nlm.nih.gov/34071832/